CLINICAL TRIAL: NCT05577832
Title: Testing Different Methods of Intramuscular Injection : A Randomized Controlled Study
Brief Title: Testing Different Methods of Intramuscular Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MusAlparlanU
Record Dates: First submitted 2022-10-05; First posted 2022-10-13 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Injection Fear; Injection Site Bruising; Pain, Acute; Satisfaction, Patient; Hematoma
MeSH Terms: conditions — Iatrophobia; Acute Pain; Patient Satisfaction; Hematoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): 3 different injection techniques in Single Group design, 1 ml intramuscular injection of dodex amp 1 ml will be applied to the deltoid muscle, one technique per week, for 1 weeks(3 day). The effects of the three techniques on pain, satisfaction with hematoma, comfort and fear of injection will be compared.
  Interventions: Procedure: Helfer Skin Tap Technique; Procedure: ShotBlocker Technique; Procedure: Standard Technique

INTERVENTIONS:
Procedure: Helfer Skin Tap Technique — In a single-group design, 3 technique injections will be administered to the patients, to be randomized. The HST technique will be applied to patients in any one of 1days in a randomized fashion.
Procedure: ShotBlocker Technique — In a single-group design, 3 technique injections will be administered to the patients, 1 technique per week, to be randomized. The ShotBlocker technique will be applied to patients in any one of 1 weeks(3 days) in a randomized manner.
Procedure: Standard Technique — Standard Technique In a single-group design, 3 technique injections will be administered to the patients, 1 technique per days, to be randomized. The standard technique will be applied to patients in any one of 1 weeks in a randomized fashion.

SUMMARY:
The goal of this clinical trial is to compare in different injection techniques. The main question[s] it aims to answer are:

* Is there a difference between the pain levels due to needle insertion in the injection made with the HST Technique, the ShotBlocker technique and the standard technique?
* Is there a difference between the hematoma levels of the injection made with the HST Technique, the ShotBlocker technique and the standard technique?
* Is there a difference between the comfort levels of the injection made with the HST Technique, ShotBlocker technique and standard technique?
* Is there a difference between the satisfaction levels of the patients with the injection made with the HST Technique, ShotBlocker technique and standard technique?
* Is there a difference between the injection fear levels of patients with HST Technique, ShotBlocker technique and standard technique?

DETAILED DESCRIPTION:
Type of Research This project is a randomized controlled trial. Place and Time of Research The research will be carried out with patients who applied to the emergency department of Atatürk University Research Hospital for IM injection between January and May 2023.

Population and Sample of the Research The population of the research will be the patients who applied to the emergency department of Atatürk University Research Hospital and were prescribed Dodex 1ml amp for IM injection. The preference of patients who were prescribed Dodex 1ml in the study is due to the fact that the treatment procedure should be administered daily, at first, and then once a week.

Dodex 1ml amp application procedure It is a red colored solution in the form of 1 ml ampoules, used in the treatment of pernicious anemia, hyperchromic macrocytic anemia, neuralgia, neuritis, sciatica, containing cyanocobalamin, that is, vitamin B12. The reason for choosing Dodex treatment is that it is a frequently used drug, it is a suitable drug (1 ml) to be applied to the deltoid region, and a certain part of the treatment is done once a week. 1 ml ampoule of Dodex In anemia due to vitamin B12 deficiency, treatment is started with 250-1000 mcg vitamin B12 4/7 application every other day and this application is continued for 1-2 weeks. Then, 250 mcg of vitamin B12 is administered once a week until the results of the blood tests prove that normalcy has returned.

Ordering the Application to the Research Group As a result of the power analysis, 40 people are planned to be included in the study. Since 3 different applications will be evaluated once a week for 1 weeks(3 day), it is planned to apply the methods to be applied to the patients in a randomized order in order to avoid bias in the research. The researcher classified the methods as A, B, C. In order to determine which methods A, B, C would be, he wrote the names of the methods on 3 pieces of paper and drew them in order. In this direction; Method A: HST Technique, Method B: Standard Technique, Method C was chosen as the Shotbocker Technique. Methods A, B, C were classified as ABC, ACB, BAC, BCA, CAB, CBA, respectively. In the same way, the researcher wrote these methods on 6 papers and drew them in order. Thus, he determined the order of methods to be applied to the patient group. ACB, BAC, CAB, BCA, CBA, ABC rankings were drawn, respectively. The order of application of the methods was determined according to the order of the patients to be included in the study.

Method A: HST Process Steps

1. Checking the physician's order.
2. Confirming the identity of the patient, the name of the drug, the dose, route and time of administration.
3. Obtaining information from the patient about his/her allergic status.
4. Checking the expiration date of the drug.
5. Ensuring hand hygiene.
6. Preparing the correct dose of the drug from the ampoule using the surgical aseptic technique.
7. Changing the needle tip
8. Patient authentication
9. Do not close the room door or pull the curtain at the bedside
10. Explaining the purpose of the treatment and the way of application to the patient before the procedure.
11. Do not wash your hands and wear disposable gloves.
12. Putting the patient in the Fowler position
13. Do not cover the patient to expose only the Deltoid region.
14. Detection of deltoid region. (In the determination of the deltoid region, a horizontal line will be drawn about one centimeter below the acromion process of the upper arm towards the outer lateral surfaces of the arm, both ends of this imaginary line will be joined at the axillary level to obtain an inverted triangle. The midpoint of the triangle shows the injection point.)
15. Cleaning around the injection site with an antiseptic tampon and in circular motions, overflowing the injection site, waiting for the area to dry.
16. Removing the needle sheath and holding the syringe between the thumb and forefinger of the active hand.
17. -Do not hit the lower part of the injection site, the lower part of the deltoid muscle twice, in a way that does not hurt the patient and does not touch the injection site. In the 3rd tapping process, penetrating the detected area with a needle to synchronize with tapping.
18. As soon as the needle is inserted, hold the lower end of the syringe using the thumb and index finger of the passive hand and check for blood by pulling back the plunger with the active hand.
19. Holding the plunger with the active hand, injecting the drug at a rate of 10 seconds/ml.
20. Wait 10 seconds before withdrawing the needle.
21. With the fourth stroke, withdraw the needle straight and steady at the angle entered into the tissue.
22. Applying light pressure to the area, without massaging, using a dry gauze or cotton pad.
23. Do not throw the needle into the sharps waste box without putting on the sheath of the used needle.
24. Gathering the materials and giving the patient a comfortable position.
25. Removing gloves and maintaining hand hygiene.
26. Saving the application.
27. Evaluating and recording the individual's response to the application. Method B: Standard Technical Application Procedure

1) Process steps 1-15 in Method A will be applied. 2) Removing the needle sheath and holding the syringe between the thumb and forefinger of the active hand.

3) As soon as the needle is inserted, hold the lower end of the syringe using the thumb and forefinger of the passive hand and check for blood by pulling back the plunger with the active hand.

4) Injecting the drug at a rate of 10 seconds/ml by holding the plunger with the active hand.

5) Wait 10 seconds before retracting the needle. 6) Straight and steady retraction of the needle with the angle inserted into the tissue.

7) Process steps 22-27 in Method A will be applied. Method C: Shotblocker Application Procedure

1. Process steps 1-15 in Method A will be applied.
2. Placing the ShotBlocker device over the deltoid region and applying light pressure on it.
3. Removing the needle sheath and holding the syringe between the thumb and forefinger of the active hand.
4. Inserting the needle into the tissue from the middle of the ShotBlocker device at an angle of 72-90 degrees.
5. As soon as the needle is inserted, hold the lower end of the syringe using the thumb and index finger of the passive hand and check for blood by pulling back the plunger with the active hand.
6. Holding the plunger with the active hand, injecting the drug at a rate of 10 seconds/ml.
7. Wait 10 seconds before retracting the needle.
8. Withdraw the needle straight and steady at the angle entered into the tissue.
9. Removing the ShotBlocker device on the deltoid region.
10. Process steps 22-27 in Method A will be applied Data Collection Before starting the research, patients will be given information about the purpose, method, etc. of the research, and the "Sociodemographic Characteristics Form" will be filled in with the patients who agree to participate in the research. Three different methods will be applied to the patients once a week. "Visual Comparison Scale", "Comfort Scale", Injection Satisfaction Evaluation Scale", "Pain Level and Duration Record Form", "Injection Fear Scale" and "Injection Application Form" will be prepared for each application separately. These forms will be filled after each application. "Opsite-Flexigrid Measurement Registration Form" will be filled in 48 hours after injection applications.

Analysis of Data The data will be evaluated in the SPSS package program. In the evaluation of the data, the statistical significance value will be accepted as 0.05, the Type 1 error will be kept at 5% and the evaluation will be made with a 95% confidence interval. In order to determine the reliability of the measurement tools, the Cronbach Alpha Value will be examined, and analyzes will continue for measurements above 0.60. Skewness and Kurtosis values will be examined in order to determine whether the measurements show a normal distribution. The data will be analyzed in the light of this information. In intra-group pre-test post-test score comparisons, the t-test for normally distributed measurements will be used for dependent samples, and the Mann-Whitney U test will be used for non-normally-distributed measurements. In order to determine the difference in repeated measurements, one-factor anova for Replicated Measurements will be used for normally distributed measurements, and Friedman test will be used for non-normally distributed measurements. In order to determine from which groups the difference originates, the t-test will be used for normally distributed measurements in dependent groups, and the Wilcoxon Ordered Signs test will be used for non-normally-distributed measurements.

Variables of the Study Independent Variable: Intramuscular injection techniques to be applied to patients (HST, Shotblocker, Standard Technique) Dependent Variables: Patients' pain levels due to needle insertion, drug-induced pain level and pain duration, hematoma frequency and levels, comfort levels, satisfaction levels, injection fear levels.

Limitations of the Research One of the limitations of the study was the inclusion of patients who were prescribed a weekly intramuscular injection of Dodex 1 ml amp.

ELIGIBILITY:
Inclusion Criteria:

1. be over 18 years old
2. Having intramuscular Dodex 1 ml amp injection treatment once a week for at least 3 consecutive weeks
3. Not using anticoagulant drugs
4. Absence of scarring, incision, lipodystrophy, infection at the injection site
5. Absence of a history of drug allergy
6. Absence of any disease that prevents perception of pain, fear and similar variables (vision, hearing, loss of sensation, cognitive disability, stroke, DM)
7. Not using centrally or peripherally effective analgesics or sedatives
8. Lack of arm limbs
9. Body mass index within normal limits
10. Prescribing Dodex amp 1 ml

Exclusion Criteria:

1. Failure to show up 3 times for injection administration
2. Drug-induced allergy development
3. The patient's desire to withdraw from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 3 days
  Patients will be asked to indicate and mark their post-injection pain, comfort, satisfaction, and fear of injection, with a minimum of 1 and a maximum of 10.
Opsite-Flexigrid Measurement Registration Form | 3 days
  The Opsite-Flexigrid Measuring Tool is an easy-to-use film cover with transparent adhesive and moisture permeability. Opsite-Flexigrid consists of a thin polyurethane membrane coated with an acrylic adhesive layer. It is used in the measurement of hematoma diameter due to its small squares and transparency. After each injection, this tape will be attached to the arm of the individual with the injection site exposed, and will be used to determine the presence of hematoma in the individual 48 hours later. It consists of squares of centimeters divided into 10 parts of 0.1mm. Hematoma sizes measured with a transparent tape will be considered as pinpoint = needle tip if a spot-shaped color change has occurred at the needle entry point, medium if it is between 0.2-1 cm2, and large hematoma if it is larger than 1 cm2. The obtained data will be recorded in the form.

CONTACTS AND LOCATIONS:
Overall Officials: Bahar Çiftçi, Study Director — Ataturk University
Locations (1):
- Atatürk University, Erzurum, Erzusum, Turkey (Türkiye)

REFERENCES:
- [Derived] Yildiz GN, Ciftci B. Deltoid muscle intramuscular injection methods examining pain comfort satisfaction and fear in ShotBlocker helfer skin tap and standard techniques. BMC Nurs. 2025 Apr 8;24(1):390. doi: 10.1186/s12912-025-02901-8. PMID 40200340